CLINICAL TRIAL: NCT03188926
Title: Surgical Treatment for Long Bone Metastases With Intramedullary Nail or Endoprosthetic Reconstruction
Brief Title: Surgical Treatment of Long Bone Metastases
Acronym: MTC
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Costantino Errani, MD, PhD, Istituto Ortopedico Rizzoli
Other Study IDs: 0026106
Record Dates: First submitted 2017-06-09; First posted 2017-06-16 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Bone Metastases; Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: intramedullary fixation or endoprosthetic reconstruction — Surgical treatment of impending or pathologic fracture in the extremities

SUMMARY:
To provide treatment guidelines for patients with long bone metastatic disease based on observational study and to propose an algorithm to guide orthopedic surgeons in decision-making for these patient.

DETAILED DESCRIPTION:
The objectives of this study were to examine clinical outcomes after reconstruction with intramedullary fixation (IMN) or endoprosthetic reconstruction (EPR) with a specific focus on (1) the rate of complication or failure; (2) differences in complication rates by anatomic site; (3) functional results as assessed by the Musculoskeletal Tumor Society System (MSTS); (4) differences in complication rate between patients treated with INM versus EPR; and (5) differences in survival in patients with metastatic bone disease based on disease-specific, laboratory, and demographic information.

ELIGIBILITY:
Inclusion Criteria:

* bone metastases of the extremity

Exclusion Criteria:

* bone metastases of the spine

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with long bone metastases treated surgically with intramedullary nail or endoprosthetic reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes after treatment of long bone metastases with intramedullary nail versus endoprosthetic reconstruction | 1 year
  The objectives of this study were to examine clinical outcomes after reconstruction with intramedullary nail versus endoprosthetic reconstruction with a specific focus on differences in complication rate between patients treated with intramedullary nail versus endoprosthetic reconstruction

SECONDARY OUTCOMES:
Survival in patients undergoing surgery for metastatic bone disease | 1 year
  Provide a reliable and objective means of estimating survival in patients with metastatic bone disease based on disease-specific

CONTACTS AND LOCATIONS:
Overall Officials: Davide Donati, MD, Study Director — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
publish a manuscript in international journal